CLINICAL TRIAL: NCT01481896
Title: A Five-Year Metal-on-Metal Retrospective Clinical Study
Status: Completed | Type: Observational
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Robert H. Hopper, Jr., Director, Anderson Orthopaedic Research Institute
Other Study IDs: AORI2011-0100; Study #09013 (Other Grant/Funding Number: DePuy Orthopaedics, Inc.)
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Results first posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis
Keywords: Hip replacement; Metal-on-metal bearings; Osteolysis; Metal ion levels; Outcome
MeSH Terms: conditions — Osteoarthritis; Osteolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metal-on-Metal Total Hip Arthroplasties: Consecutive series of patients who had metal-on-metal primary total hip arthroplasty performed with DePuy Pinnacle cups, Ultamet metal liners and 36-mm cobalt-chromium alloy femoral heads.
  Interventions: Device: Metal-on-metal primary total hip arthroplasty (DePuy )

INTERVENTIONS:
Device: Metal-on-metal primary total hip arthroplasty (DePuy ) — Replacement of a patient's native hip with an artificial implant featuring a metal-on-metal articulation
  Other Names: DePuy Pinnacle acetabular cup; DePuy Ultamet metal liner; DePuy 36-mm femoral head

SUMMARY:
This retrospective study will review the Anderson Orthopaedic Institute's initial experience among a consecutive series of 126 patients who had primary total hip arthroplasty using a metal-on-metal articulation consisting of a DePuy Pinnacle cup with an Ultamet liner coupled with a 36-mm cobalt-chrome alloy femoral head. The relationship between metal ion levels, cup orientation, osteolysis, radiographic implant stability and clinical outcome measures including component revision, complications, patient satisfaction and Harris Hip Scores will be evaluated.

DETAILED DESCRIPTION:
Metal-on-metal bearings for total hip arthroplasty are an alternative to traditional polyethylene bearing surfaces and hip simulators studies have shown that metal-on-metal bearings have lower wear than metal-on-polyethylene bearings. In addition, simulator studies indicate that the amount of wear decreases as head size increases allowing the use of larger head diameters than possible with other bearing surfaces. Since dislocation is currently the most common reason for reoperation in the United States, representing 22.5% of hip revisions, the combination of low wear and larger head sizes to reduce dislocation hold the promise of improving outcome among total hip arthroplasty patients. While there are potential advantages to metal-on-metal bearings, a few concerns have been noted in the literature. Although the total volume of wear is low with these bearings, the articulation generates metal debris that may be related to patient and surgical factors such as implant positioning. Despite a reduced wear volume, there is also the possibility that an increased bioreactivity associated with metal debris might induce an osteolytic response or local tissue hypersensitivity reaction.

This study will retrospectively review the outcome of a consecutive series of 126 patients who had 131 primary THAs performed between April 2001 and November 2002 at the Anderson Clinic with a Pinnacle acetabular cup, an Ultamet insert and a 36-mm cobalt-chrome alloy femoral head. These total hip arthroplasties represent the Anderson Orthopaedic Institute's in initial experience with this implant. The relationship between metal ion levels, cup orientation, osteolysis, radiographic implant stability and clinical outcome measures including component revision, complications, patient satisfaction and Harris Hip Scores will be evaluated. The outcome data from our analysis will also be compared with the data from other published series with metal-on-metal bearing surfaces. Serial radiographs obtained as part of routine post-operative care will be used to evaluate osteolysis, implant stability and radiographic complications such as periprosthetic fracture. The area of each osteolytic region will be measured on the AP pelvic x-ray using Martell's Hip Analysis Suite. Computed tomography (CT) scans obtained as part of routine follow-up will be also analyzed to identify regions of acetabular osteolysis. The volume and location of each osteolytic defect identified on CT will be evaluated using three-dimensional image analysis software (Analyze, Biomedical Imaging Resource, Rochester, MN). A three-dimensional (3D) reconstruction of the pelvis, cup and acetabular osteolytic lesions will also be generated from the CT image data. This reconstruction will be oriented to simulate the AP pelvic radiographic view. Cobalt and chromium ion level data will be compiled for patients who had blood drawn to evaluate metal ion levels. The mean and median blood metal-ion levels for these patients will be calculated and the results will be compared to the metal-ion levels reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty patients who had surgery between April 2001 and November 2002 who were implanted with a Pinnacle acetabular cup, an Ultamet metal-on-metal insert and a 36mm cobalt-chrome alloy femoral head

Exclusion Criteria:

* Revision total hip arthroplasties
* Primary total hip arthroplasties using Ultamet liners coupled with 28-mm femoral heads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients who had primary total hip arthroplasties performed at the Anderson Clinic using DePuy Pinnacle cups, Ultamet metal liners and 36-mm cobalt-chromium alloy femoral heads.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hopper, Jr., PhD, Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

REFERENCES:
- [Background] MacDonald SJ. Metal-on-metal total hip arthroplasty: the concerns. Clin Orthop Relat Res. 2004 Dec;(429):86-93. doi: 10.1097/01.blo.0000150309.48474.8b. PMID 15577471
- [Background] Bozic KJ, Kurtz S, Lau E, Ong K, Chiu V, Vail TP, Rubash HE, Berry DJ. The epidemiology of bearing surface usage in total hip arthroplasty in the United States. J Bone Joint Surg Am. 2009 Jul;91(7):1614-20. doi: 10.2106/JBJS.H.01220. PMID 19571083
- [Background] Bozic KJ, Kurtz SM, Lau E, Ong K, Chiu V, Vail TP, Rubash HE, Berry DJ. The epidemiology of revision total knee arthroplasty in the United States. Clin Orthop Relat Res. 2010 Jan;468(1):45-51. doi: 10.1007/s11999-009-0945-0. Epub 2009 Jun 25. PMID 19554385
- [Background] Dowson D, Hardaker C, Flett M, Isaac GH. A hip joint simulator study of the performance of metal-on-metal joints: Part II: design. J Arthroplasty. 2004 Dec;19(8 Suppl 3):124-30. doi: 10.1016/j.arth.2004.09.016. PMID 15578566
- [Background] Rieker CB, Schon R, Kottig P. Development and validation of a second-generation metal-on-metal bearing: laboratory studies and analysis of retrievals. J Arthroplasty. 2004 Dec;19(8 Suppl 3):5-11. doi: 10.1016/j.arth.2004.09.017. PMID 15578545
- [Background] Silva M, Heisel C, Schmalzried TP. Metal-on-metal total hip replacement. Clin Orthop Relat Res. 2005 Jan;(430):53-61. doi: 10.1097/01.blo.0000149995.84350.d7. PMID 15662304
- [Background] Beaule PE, Campbell P, Mirra J, Hooper JC, Schmalzried TP. Osteolysis in a cementless, second generation metal-on-metal hip replacement. Clin Orthop Relat Res. 2001 May;(386):159-65. doi: 10.1097/00003086-200105000-00020. PMID 11347829
- [Background] Willert HG, Buchhorn GH, Fayyazi A, Flury R, Windler M, Koster G, Lohmann CH. Metal-on-metal bearings and hypersensitivity in patients with artificial hip joints. A clinical and histomorphological study. J Bone Joint Surg Am. 2005 Jan;87(1):28-36. doi: 10.2106/JBJS.A.02039pp. PMID 15637030
- [Background] Engh CA Jr, Ho H, Engh CA. Metal-on-metal hip arthroplasty: does early clinical outcome justify the chance of an adverse local tissue reaction? Clin Orthop Relat Res. 2010 Feb;468(2):406-12. doi: 10.1007/s11999-009-1063-8. Epub 2009 Sep 1. PMID 19727991
- See also: Website for Anderson Orthopaedic Research Institute — http://aori.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this retrospective study, the Anderson Orthopaedic Research Institute's database was used to identify a consecutive series of the first 126 patients who had 131 primary total hip arthroplasties using a Pinnacle acetabular cup, an Ultamet metal-on-metal insert and a 36-mm cobalt-chrome alloy femoral head.
Pre-assignment Details: No patient from the consecutive series of hip replacements performed between April 2001 and November 2002 was excluded.
Groups:
- Metal-on-Metal Total Hip Arthroplasties: Consecutive series of primary total hip arthroplasties performed with DePuy Pinnacle cups, Ultamet metal liners and 36-mm cobalt-chromium alloy femoral heads.
Period: Overall Study
Arm/Group | Metal-on-Metal Total Hip Arthroplasties
Started | 126 (The 126 participants includes 5 participants with bilateral hip replacements for a total of 131 THAs)
Min 4.75 yr Follow-up, Revised or Dead | 114 (114 participants with 119 THAs had at least 4.75 year follow-up or were known revised or deceased)
Completed | 114 (The 114 participants includes 5 participants with bilateral hip replacements for a total of 119 THAs)
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants is defined as the number of hips included in the study population instead of the number of participants since 5 participants had both hips replaced and objective of this study was to evaluated the outcome of each hip.
Arm/Group | Metal-on-Metal Total Hip Arthroplasties
Number analyzed (Participants) | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 121
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 74
Region of Enrollment [Number; unit: participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Metal Ion Levels Per Participant
Description: Metal ion levels include cobalt and chromium ion levels determined from tests of blood samples. Metal ion levels are reported per participant since blood samples were taken from individual participants who could have had one or both hips replaced.
Time Frame: At a mean of 4.2 years after primary total hip arthroplasty
Population: Patients who had blood drawn and analyzed for serum cobalt levels as part of routine care are included.
Measure: Median (Full Range); unit: micrograms per liter
Groups:
- Patients With Serum Cobalt Levels: Patients were recommended to have blood drawn for evaluation of serum cobalt levels if they were considered to be active or thought to be at risk for an adverse local tissue reaction. Blood was drawn at our hospital or a facility of the patient's choice. Among all the labs that performed metal level assessments, the cobalt detection limit varied from 0.5 to 1.0 microgram per liter. Patients with undetectable cobalt levels were assigned a value of zero. A patient's cobalt level was considered high if it was 7 micrograms per liter or greater.
- Patients With Serum Chromium Levels: Patients were recommended to have blood drawn for evaluation of serum chromium levels if they were considered to be active or thought to be at risk for an adverse local tissue reaction. Blood was drawn at our hospital or a facility of the patient's choice. The chromium detection limit was 0.1 micrograms per liter for all labs that performed metal level assessments. Patients with undetectable chromium levels were assigned a value of zero. A patient's chromium level was considered high if it was 7 micrograms per liter or greater.
Arm/Group | Patients With Serum Cobalt Levels | Patients With Serum Chromium Levels
Number analyzed (Participants) | 65 | 62
micrograms per liter | 1.4 [0 to 37] | 2.1 [0 to 28.9]

2. Secondary Outcome: Cup Orientation Per Hip
Description: Cup orientation including abduction and anteversion is determined using follow-up radiographs. Since a participant with both hips replaced could have different cup orientations for each hip, cup abduction and anteversion angles are reported per hip.
Time Frame: On the first post-operative anteroposterior pelvic radiograph after primary total hip arthroplasty
Population: Cup orientation was measured for all 131 total hip replacements included in the study population.
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: hips
Groups:
- Cup Abduction Angle: The Cup Abduction Angle quantifies the amount of tilt associated with the hemispheric implant implanted inside a patient's pelvis to replace their hip socket. When an anterioposterior (front-to-back) x-ray is taken, the angle between the face of the cup and a horizontal line defines the Cup Abduction Angle. The line defining the face of the cup is drawn through the uppermost and lowest edges of the cup's projection on the x-ray. For this study, the Cup Abduction Angle was measured from digitized x-rays using Dr. John Martell's Hip Suite Analysis Software (University of Chicago, Chicago, IL).
- Cup Anteversion Angle: The Cup Anteversion Angle quantifies the front-to-back rotation of the hemispheric implant implanted inside a patient's pelvis to replace their hip socket. When an anterioposterior (front-to-back) x-ray is taken, the circular face of the cup projects onto the x-ray as an ellipse. The ratio of the major axis of the ellipse to the minor axis can be used to calculate the anteversion. A cup rotated anteriorly has positive anteversion. A cup rotated posteriorly has negative anteversion. For this study, the cup Anteversion Angle was measured from digitized x-rays using Dr. John Martell's Hip Suite Analysis Software (University of Chicago, Chicago, IL). Taken together, the abduction and anteversion angle quantify the three-dimensional orientation of the cup.
Arm/Group | Cup Abduction Angle | Cup Anteversion Angle
Number analyzed (Participants) | 126 | 126
Number analyzed (hips) | 131 | 131
degrees | 39 [23 to 59] | 19 [7 to 35]

3. Secondary Outcome: Harris Hip Score Per Hip
Description: Harris Hip Scores are derived from a patient questionnaire and physical examination. Since a participant with both hips replaced could have different Harris Hip Scores for each hip, the Harris Hip Scores are reported per hip.
Time Frame: At a mean of 5.6 years after primary total hip arthroplasty
Measure: Median (Full Range); unit: units on a scale
Units Other Than Participants: hips
Groups:
- Hips With Harris Hip Scores: The Harris Hip Score is an outcome measure used for hip replacements that ranges from 0 (worst) to 100 (best). The score consists of a series of questions related to hip pain, function and range of motion that accumulate a different number of points depending on the response choices. At the time of their follow-up visits, patients completed a standardized questionnaire that included components of the Harris Hip Score and the physician completed a standardized evaluation which included range of motion assessment.
Arm/Group | Hips With Harris Hip Scores
Number analyzed (Participants) | 110
Number analyzed (hips) | 114
units on a scale | 95 [49 to 100]

4. Secondary Outcome: Osteolysis Per Hip
Description: Osteolysis is defined as localized areas of peri-prosthetic bone loss that did not exist prior to surgery and is evaluated using radiographs and CT scans. Since a participant with both hips replaced could have a osteolysis present or absent for each hip, osteolysis is reported per hip.
Time Frame: At a mean of 5.6 years after primary total hip arthroplasty
Population: Patients who had radiographs or computed tomography (CT) scans taken as part of routine care were included.
Measure: Number; unit: Number of hips with osteolysis
Units Other Than Participants: hips
Groups:
- Hips With Radiographs Analyzed for Femoral Osteolysis: Serial x-rays for each hip replacement were analyzed by a single experienced reviewer to identify regions where bone had been lost in the femur. Expansile (ballooned-out) regions of bone loss identified on follow-up x-rays taken at least 4.75 years after their surgery that were not apparent on the immediate post-operative x-ray were considered to be osteolysis. For the purposes of reporting, the total number of hips with any evidence of femoral osteolysis on x-ray is indicated.
- Hips With CT Scans Analyzed for Pelvic Osteolysis: Digital Computed Tomography (CT) scans taken more than 5 years after a patient's hip replacement were used to evaluate pelvic bone loss (osteolysis). Regions of bone loss were traced on CT slices to determine the volume and location of each osteolytic defect using three-dimensional image analysis software (Analyze, Biomedical Imaging Resource, Rochester, MN). For the purposes of reporting, the total number of hips with any evidence of pelvic osteolysis on CT is indicated.
Arm/Group | Hips With Radiographs Analyzed for Femoral Osteolysis | Hips With CT Scans Analyzed for Pelvic Osteolysis
Number analyzed (Participants) | 104 | 35
Number analyzed (hips) | 108 | 38
Number of hips with osteolysis | 3 | 2

5. Secondary Outcome: Implant Stability Per Hip
Description: Implant stability is classified and stable/bone ingrown, fibrous fixed or loose and evaluated using conventional radiographs. Since a participant with both hips replaced could have a different type of stability for each hip, implant stability is reported per hip.
Time Frame: At a mean of 5.6 years after primary total hip arthroplasty
Population: All hips that had a follow-up x-ray taken at least 4.75 years after their joint replacement were included.
Measure: Number; unit: number of hips
Units Other Than Participants: hips
Groups:
- Stem Stability: Based on the most recent follow-up x-ray, the fixation of the stem component implanted in a patient's femur was graded as bone ingrown, fibrous stable or loose using the criteria defined by Engh, Massin and Suthers in their article titled "Roentgenographic assessment of the biologic fixation of porous-surfaced femoral components" published in the August 1990 edition of Clinical Orthopaedics and Related Research on pages 107 to 128.
- Cup Stability: Based on the most recent follow-up x-ray, the fixation of the cup component implanted in a patient's pelvis was graded as bone ingrown, fibrous stable or loose. A cup was considered fibrous stable if there was a continuous radiolucent line along the interface between the cup and the patient's pelvic bone. A cup was considered loose if it had migrated more than 2 mm or its orientation had changed by at least 5 degrees on the follow-up x-ray compared to the immediate post-operative x-ray. A cup that did not meet the criteria for fibrous stable or loose was considered bone ingrown.
Arm/Group | Stem Stability | Cup Stability
Number analyzed (Participants) | 104 | 104
Number analyzed (hips) | 108 | 108
number of hips
  Bone ingrown | 105 | 108
  Fibrous stable | 2 | 0
  Loose | 1 | 0

6. Secondary Outcome: Component Revision Per Hip
Description: For implants that require a component revision, the reason for the revision is determined based on the pre-operative history and operative findings at the time of revision. Since a participant with both hips replaced could have a revision of each hip, component revision is reported per hip.
Time Frame: At a mean of 6.7 years after primary total hip arthroplasty
Measure: Number; unit: number of hips
Units Other Than Participants: hips
Arm/Group | Metal-on-Metal Total Hip Arthroplasties
Number analyzed (Participants) | 126
Number analyzed (hips) | 131
number of hips
  Stem revision for aseptic loosening | 1
  Broken stem | 2
  Liner & head exchange for groin pain & osteolysis | 1

7. Secondary Outcome: Patient Satisfaction Per Hip
Description: Whether or not an individual is satisfied with the outcome of their hip arthroplasty is evaluated using a questionnaire. Since a participant with both hips replaced could have a different level of satisfaction for each hip, patient satisfaction is reported per hip.
Time Frame: At a mean of 5.6 years after primary total hip arthroplasty
Measure: Number; unit: number of participants
Units Other Than Participants: hips
Groups:
- Patients Satisfied With Outcome of Hip Replacement: Patient satisfaction was evaluated by asking the question, "Are you satisfied with the results of your hip operation?" on a questionnaire. Patients could respond "Yes" or "No" by filling in the appropriated bubble on the questionnaire.
Arm/Group | Patients Satisfied With Outcome of Hip Replacement
Number analyzed (Participants) | 102
Number analyzed (hips) | 106
number of participants
  Satisfied | 106
  Unsatisfied | 0

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from the time of surgery to a mean follow-up of 6.7±2.4 years, ranging from 0 to 10.8 years, and were compiled by querying the Anderson Orthopaedic Research Institute's database for post-operative complications and revisions.
Description: All 131 hips were considered at risk for each of the adverse events with the following exceptions: death uses the 126 study participants; elevated ion levels uses the 65 patients with ion measurements; femoral osteolysis, stem loosening and fibrous stem stability use the 108 hips with x-rays; and pelvic osteolysis uses the 38 hips with CT scans.
Arm/Group | Metal-on-Metal Total Hip Arthroplasties
Serious Adverse Events (participants affected / at risk) | 12/131
Other Adverse Events (participants affected / at risk) | 16/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Metal-on-Metal Total Hip Arthroplasties (N=131)
Component Revision (Surgical and medical procedures) | 4 (4) — Loose stem revised at 3.0 years; Broken stem revised at 4.6 years; Metal liner & head revised at 8.5 years for femoral osteolysis, groin pain, metallosis and implant corrosion; Broken stem with metal liner & head revised at 9.6 years with corrosion
Death (General disorders) | 4/126 (4) — Patients died 3 days, 6.5 years, 7.8 years and 8.0 years after their hip replacements at ages of 77.3, 53.9, 82.0 and 72.2 respectively. Death at 3 days thought to be due to a sudden cardiac event.
Irrigation & Debridement for Hematoma (Surgical and medical procedures) | 1 (1) — After a hip aspiration to rule out infection 12 days post-operatively, patient presented with severe pain 14 days post-operatively and approximately 500 cc of dense hematoma was removed during a hip exploration.
Irrigation & Debridement for Infection (Surgical and medical procedures) | 1 (1) — Patient presented with increasing pain, fever and a wound that had begun to drain slightly serous fluid. An incision and drainage for acute infection was performed 0.05 years post-operatively. Intra-operatively cultures grew Staphylococcus aureus.
Dislocation (Surgical and medical procedures) | 1 (1) — Patient sustained a dislocation 5.5 years post-operatively that was reduced in the Emergency Room.
Post-operative Fat Embolism (Vascular disorders) | 1 (1) — Patient developed a decrease in metal status along with hypoxia and decreased blood pressure during the evening after surgery and was thought to have had a fat embolism or a reaction to post-operative medications.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Metal-on-Metal Total Hip Arthroplasties (N=131)
Serum Metal Levels of 7 micrograms/L or higher (Blood and lymphatic system disorders) | 6/65 (6) — At a mean follow-up of 4.5 years (range 1.0-6.3), 6 patients had cobalt or chromium levels of at least 7 based on results from community labs. Among these 6, median cobalt level was 26 (range 4.8-37) and median chromium level was 7.4 (range 2.9-28.9)
Femoral osteolysis on x-ray (Musculoskeletal and connective tissue disorders) | 3/108 (3) — Three patients had osteolysis confined to the proximal femur that was identified on routine follow-up x-rays taken at 5.0, 5.5, and 5.6-year follow-up.
Pelvic osteolysis on computed tomography scan (Musculoskeletal and connective tissue disorders) | 2/38 (2) — Two patients had pelvic osteolysis identified at the cup rim on computed tomography scans. One had a 2.7 cubic centimeter inferior rim defect at 5.1 year follow-up. The other had 7.4 cubic centimeter anterior rim defect at 5.2 year follow-up.
Loose stem on x-ray (Musculoskeletal and connective tissue disorders) | 1/108 (1) — A loose stem was identified on a routine follow-up x-ray taken at 5.1-year follow-up.
Hip Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient reported a subluxation that occurred 2.6 years post-operatively and self-reduced.
Greater Trochanter Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) — One patient had an asymptomatic fracture on a 6-week follow-up radiograph that was not treated. Another patient sustained a non-displaced fracture 8.0 years post-operatively secondary to a bicycle accident that also resulted in other injuries.
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient presented with right groin pain 0.4 years post-operatively and was diagnosed with iliopsoas tendonitis.
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient reported intermittent thigh pain at 8.6 year follow-up that began about 2 years previously.
Pubic ramus fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient sustained a pubic ramus fracture 5.4 years post-operatively that healed without intervention.
Abnornal sensation with range of motion (Musculoskeletal and connective tissue disorders) | 1 (1) — At a routine follow-up appointment 1.1 years post-operatively, patient reported that hip seemed to "grab" in certain positions.
Fibrous stable stem (Musculoskeletal and connective tissue disorders) | 2/108 (2) — Two patients were noted to have fibrous stable stems that were not bone ingrown on radiographs that were obtained 5.3 years post-operatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any paper drafted regarding the results of the study shall be sent to Depuy Clinical Research for review and comment at least thirty (30) days before being submitted for publication; the same shall apply to abstracts, except the time for review by DePuy shall be ten (10) days. DePuy will promptly inform the authors of any changes deemed necessary to preserve the confidentiality of proprietary information or to ensure scientific accuracy.